CLINICAL TRIAL: NCT06836232
Title: A Phase 2a, Open-Label Pilot Study to Evaluate the Safety/Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of VTX2735 in Participants With Recurrent Pericarditis
Brief Title: An Open-Label Pilot Study of VTX2735 in Recurrent Pericarditis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zomagen Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTX2735-202
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Pericarditis
Keywords: Ventyx; Zomagen; Recurrent Pericarditis; VTX2735; NLRP3 Inhibitor; NLRP3; Inflammasome
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental)
  Interventions: Drug: VTX2735
- Cohort B Treatment Group B1 (Experimental)
  Interventions: Drug: VTX2735
- Cohort B Treatment Group B2 (Experimental)
  Interventions: Drug: VTX2735

INTERVENTIONS:
Drug: VTX2735 — Dose A, daily
  Arms: Cohort A
Drug: VTX2735 — Dose B, Daily
  Arms: Cohort A; Cohort B Treatment Group B1
Drug: VTX2735 — Dose C, daily
  Arms: Cohort B Treatment Group B2

SUMMARY:
This is a study to understand if taking VTX2735 is safe and effective in participants diagnosed with Recurrent Pericarditis (RP).

Cohort A will include up to 30 participants and will consist of the following:

* A 30-day Screening Period (to see if a participant qualifies for the study)
* A 6-week Open Label Treatment Period - participant receives VTX2735 Dose A
* A 7-week Extension Treatment Period (if a participant meets criteria for extension treatment) - participant receives VTX2735 Dose A
* An 11-week Once Daily Treatment Period (if a participant meets criteria for this treatment period) - participant receives VTX2735 Dose B
* A 14-day Follow-Up Period

Cohort B will include up to 20 participants and will consist of the following:

* A 30-day Screening Period (to see if a participant qualifies for the study)
* A 6-week Open Label Treatment Period - participant receives VTX2735 Dose B or C
* An 18-week Extension Treatment Period (if a participant meets criteria for extension treatment) - participant receives VTX2735 Dose B or C
* A 14-day Follow-Up Period

ELIGIBILITY:
Inclusion Criteria:

* Participants are male or female ≥ 18 years up to ≤ 75 years of age.
* Capable of giving signed informed consent and able to comply with the protocol
* Previously had an index (first) episode of pericarditis which met the criteria for an acute pericarditis event
* Ongoing symptomatic episode of pericarditis, or may have an episode of recurrent pericarditis in the next 4 weeks.
* CRP by local laboratory assessment prior to first dose of study treatment (participants with CRP ≤ 10 mg/L must be receiving corticosteroid treatment for RP and have evidence of pericardial inflammation)
* Pericarditis pain score ≥ 4 based on the 11-point NRS.
* Stable doses of NSAIDs, colchicine, and/or oral corticosteroids (if receiving these treatments)

Exclusion Criteria:

* Current or prior diagnosis of pericarditis that is secondary to specific prohibited causes, including but not limited to tuberculosis, blunt trauma, tumor, myocarditis, or systemic autoimmune diseases.
* History of clinically significant immunosuppressive disorder, autoimmune/autoinflammatory disorder, or primary or secondary immunodeficiency.
* Clinically important history of a medical disorder that would compromise safety or data quality, per the Investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of VTX2735 | Day 1 of treatment period through study completion, up to 26 weeks
  Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to study treatment discontinuation

SECONDARY OUTCOMES:
Effect of VTX2735 on pericardial pain | Day 1 of treatment period to Week 6 of treatment period
  Change from baseline in Numeric Pain Rating Scale (NRS) over time through Week 6
Effect of VTX2735 on inflammation | Day 1 of treatment period to Week 6 of treatment period
  Change from baseline in High-Sensitivity C-Reactive Protein (hs-CRP) over time through Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Sonnergren, MD, PhD, Study Director — Ventyx Biosciences
Locations (16):
- United States (16):
  - Local Site #840012, Tucson, Arizona
  - Local Site #840014, Orange, California
  - Local Site #840016, Saint Augustine, Florida
  - Local Site #840008, Chicago, Illinois
  - Local Site #840002, Park Ridge, Illinois
  - Local Site #840011, Owensboro, Kentucky
  - Local Site #840010, Boston, Massachusetts
  - Local Site #840005, Rochester, Minnesota
  - Local Site #840020, New York, New York
  - Local Site #840017, Cleveland, Ohio
  - Local Site #840019, Houston, Texas
  - Local Site #840001, Houston, Texas
  - Local Site #840013, Salt Lake City, Utah
  - Local Site #840018, Charlottesville, Virginia
  - Local Site #840004, Richmond, Virginia
  - Local Site #840021, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided